CLINICAL TRIAL: NCT04134546
Title: Early Versus Late Intervention After Biliary Tract Injury Post Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bassem Barghoth Sabet Amin, resident doctor at general surgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: biliary tract injury
Record Dates: First submitted 2019-10-10; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Biliary Fistula
MeSH Terms: conditions — Biliary Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group with biliary injury (Experimental): group for Early versus late intervention after biliary tract injury post cholecystectomy
  Interventions: Procedure: CBD exoloration

INTERVENTIONS:
Procedure: CBD exoloration — Early versus late intervention after biliary tract injury post cholecystectomy

SUMMARY:
Bile duct injury following cholecystectomy is an iatrogenic catastrophe associated with significant peri operative morbidity and mortality(1, 2) reduced long term survival(3) and quality of life(4, 5) and high rates of subsequent litigation6. It should be regarded as preventable.

The advent of laparoscopic cholecystectomy has resulted in a resurgence of interest in bile duct injury and its subsequent management. Population based studies(6.7) suggest a significant increase in the incidence of injury (0•1 to 0•5 per cent) following the implementation of the laparoscopic approach(8) Bile duct injury should be regarded as preventable, but over 70 per cent of surgeons regard it as unavoidable(9). Although most injuries occur within the surgeon's first 100 laparoscopic cholecystectomies, one third happen after the surgeon has performed more than 200; it is more than inexperience that leads to bile duct injury(10). It has been suggested that the commonest cause of common bile duct injury is misidentification of biliary anatomy (70-80 per cent of injuries)(11,12),a reduction in risk if surgeons perform routine intraoperative cholangiography Recognition of bile duct injury at the time of cholecystectomy allows an opportunity for the hepatobiliary surgeon to assess its severity and the presence of any vascular injury

DETAILED DESCRIPTION:
Bile duct injury following cholecystectomy is an iatrogenic catastrophe associated with significant peri operative morbidity and mortality(1, 2) reduced long term survival(3) and quality of life(4, 5) and high rates of subsequent litigation6. It should be regarded as preventable.

The advent of laparoscopic cholecystectomy has resulted in a resurgence of interest in bile duct injury and its subsequent management. Population based studies(6.7) suggest a significant increase in the incidence of injury (0•1 to 0•5 per cent) following the implementation of the laparoscopic approach(8) Bile duct injury should be regarded as preventable, but over 70 per cent of surgeons regard it as unavoidable(9). Although most injuries occur within the surgeon's first 100 laparoscopic cholecystectomies, one third happen after the surgeon has performed more than 200; it is more than inexperience that leads to bile duct injury(10). It has been suggested that the commonest cause of common bile duct injury is misidentification of biliary anatomy (70-80 per cent of injuries)(11,12),a reduction in risk if surgeons perform routine intraoperative cholangiography Recognition of bile duct injury at the time of cholecystectomy allows an opportunity for the hepatobiliary surgeon to assess its severity and the presence of any vascular injury

ELIGIBILITY:
Inclusion Criteria:

* All patients with post cholecystectomy biliary tract injury admitted at Assuit university hospital at the period of the study

Exclusion Criteria:

* Any case with biliary leakage not post cholecystectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
faliure of interventon | two months
  By mesurment liver functon as direct billirubin

SECONDARY OUTCOMES:
plan for improving | two months
  by mesurment of liver function as AST